CLINICAL TRIAL: NCT02965612
Title: Tolerability and Side Effects for a New Device in Specific Immunotherapy for Allergic Child
Brief Title: Specific Immunotherapy for Allergic Child
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mariella Enoc (Other)
Collaborators: Bial Aristegui Italia srl (Unknown); OPBG Contract and Research Organization (Unknown)
Responsible Party: Sponsor-Investigator, Mariella Enoc, President, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 947_OPBG_2014
Record Dates: First submitted 2016-11-08; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Rhinitis; Allergic Asthma; Grass Allergy
Keywords: Grass Allergy; Allergic Rhinitis; Allergic Asthma; Paediatric
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITS with Injex (Experimental): For Each patient, at each monthly vaccination session and randomly in alternate mode, will be administered two vaccine doses of 0.25 ml each at 20 minutes from one another in the two arms, in an alternating manner via Injex and via subcutaneous.
  Interventions: Device: Injex
- SCIT: ITS via subcutaneous (Active Comparator): For Each patient, at each monthly vaccination session and randomly in alternate mode, will be administered two vaccine doses of 0.25 ml each at 20 minutes from one another in the two arms, in an alternating manner via Injex and via subcutaneous.
  Interventions: Procedure: SCIT

INTERVENTIONS:
Device: Injex — administration of Specific Immunotherapy (ITS) with car pressure injector without a needle
  Arms: ITS with Injex
Procedure: SCIT — administration of Specific Immunotherapy (ITS) via traditional subcutaneous
  Arms: SCIT: ITS via subcutaneous

SUMMARY:
The recent interest that the Specific Immunotherapy (ITS) has aroused is due to the positive potential role that could be played, in particular in the forms of allergic asthma, because this method constitute the only intervention (unlike that pharmacologic) able to act on the same causes of the disease, altering the natural history. To achieve this the investigator has tried to use the specific subcutaneous immunotherapy (SCIT), to which there are studies that, with scientific rigor, have demonstrated the benefits.

DETAILED DESCRIPTION:
The Investigator proposes to compare, in children with allergic rhinitis and / or allergic asthma to grasses, the pain caused by the administration of the Specific Immunotherapy (ITS) via epicutaneous with autoinjector (INJEX) pressure without needle vs. the traditional subcutaneous immunotherapy (SCIT).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from both parents / legal guardian;
* Of both sexes;
* Between the ages of 5 to 18 sensitized to grasses Awareness for grasses will be established with prick test;
* Rhinitis established according to the ARIA (Allergic Rhinitis and its Impact on Asthma) guidelines and / or stage 1 or 2 Asthma according to GINA classification (Global Initiative for Asthma)
* It may, or not, be going on ITS with s.c. administration

Exclusion Criteria:

* Children under age 5 and age> 18 years;
* Autoimmune diseases and immunodeficiencies;
* Neoplasms;
* Severe psychological problems;
* Treatment with β-blockers;
* Poor compliance, including language training;
* Severe asthma uncontrolled by medication or irreversible airway obstruction (FEV1 less than 70% of the predicted value);
* Severe cardiovascular diseases in which may be hazardous in the administration of adrenaline

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of pain | monthly for 6 month
  questionnaire of the pain scale monthly at each seat vaccination soon after every administration : the Wong-Baker scale for children aged 3 to 8 years and the classical analogue scale from 8 years and 1 day to 18 years.

SECONDARY OUTCOMES:
prevalence of pain | 20 minutes after every administration
  questionnaire of the pain scale monthly at each seat vaccination: the Wong-Baker scale for children aged 3 to 8 years and the classical analogue scale from 8 years and 1 day to 18 years.
Incidence of procedure adverse events | within 24-48 hours after every administration
  adverse events related to the different procedure used for the administration of the specific immunotherapy
Incidence of procedure adverse events | 6 month
  adverse event related to the different procedure used for the administration of the specific immunotherapy recorded by the patient on a special diary

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Fiocchi, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Operating unit of Allergology, Rome, Italy

IPD SHARING:
Plan to Share IPD: No